CLINICAL TRIAL: NCT03400618
Title: The Effect of Carbohydrate Content in the Diet on Mean Glucose Levels in Type 1 Diabetes
Brief Title: Carbohydrate Content in the Diet in Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Carbohydrate study
Record Dates: First submitted 2018-01-05; First posted 2018-01-17 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Carbohydrates; Diet; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate carbohydrate diet (Experimental): A healthy diet containing 30 E % carbohydrates
  Interventions: Other: Moderate carbohydrate diet
- Higher carbohydrate diet (Experimental): A healthy diet containing 50 E % carbohydrates
  Interventions: Other: Higher carbohydrate diet

INTERVENTIONS:
Other: Moderate carbohydrate diet — 30 E % carbohydrates included in the diet
  Arms: Moderate carbohydrate diet
Other: Higher carbohydrate diet — 50 E % carbohydrates included in the diet
  Arms: Higher carbohydrate diet

SUMMARY:
The aim of this study is to analyse the effect of a diet with a moderate amount of carbohydrates and compare it with a traditional diabetic diet with a higher content of carbohydrates on mean glucose level, high and low glucose levels, and the risk of ketoacidosis in patients with type 1 diabetes. The glucose levels will be measured by blinded continuous glucose monitoring (CGM).

The trial has a cross-over design and 12 weeks in duration, where patients will be randomized to; 1) a diet with moderate carbohydrate content for 4 weeks and 2) a traditional diabetes diet for 4 weeks and with a wash-out period between for 4 weeks. The two diets will both be healthy and planned by a dietitian. There will be 50 subjects included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Adults 18 years or older
* Written Informed Consent
* HbA1c ≥ 58 mmol/mol (7,5 % DCCT standard)

Exclusion Criteria:

* Pregnancy or planned pregnancy for the study duration
* Severe cognitive dysfunction or other disease, which is judged by the physician to be not suitable for inclusion
* Problems with compliance to the intervention diets (excluding a lot of the foods that are common in the diets like wholegrain/beans/lentils/fruit/vegetables) because of personal preferences, other diseases, stomach problems etc.
* Diabetes duration < 1 year
* Planned change in diabetes treatment (eg. Start with insulin pump, CGM etc.) during the study period
* Other investigator-determined criteria unsuitable for patient participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The difference in mean glucose level | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12

SECONDARY OUTCOMES:
The difference in standard deviation of glucose levels | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12
The difference in the proportion of time with high glucose levels | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12
The difference in the proportion of time with euglycaemic levels | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12
Weight | Week 4, week 12
  The difference in weight between week 4 and week 12
Total cholesterol | Week 4, week 12
  The difference in total cholesterol between week 4 and week 12
LDL cholesterol | Week 4, week 12
  The difference in LDL cholesterol between week 4 and week 12
HDL cholesterol | Week 4, week 12
  The difference in HDL cholesterol between week 4 and week 12
Triglycerides | Week 4, week 12
  The difference in triglycerides between week 4 and week 12
Total insulin dose | Week 1-4, week 9-12
  The difference in total insulin dose between week 1-4 and week 9-12
Diabetes Treatment Satisfaction Questionnaire (DTSQc) score | Week 12
  The difference in DTSQc score at week 12
Diabetes Treatment Satisfaction Questionnaire (DTSQs) score | Week 4, week 12
  The difference in DTSQs scores between week 4 and week 12
Hypoglycemia confidence score | Week 4, week 12
  The difference in hypoglycaemia confidence scores between week 4 and week 12

OTHER OUTCOMES:
The difference in Mean Amplitude of Glycemic Excursions (MAGE) | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12
HbA1c | Week 4, week 12
  The difference in HbA1c between week 4 and week 12
Apolipoproteins | Week 4, week 12
  The difference in apolipoproteins between week 4 and week 12
The difference in the proportion of time with low glucose levels | Week 3-4, week 11-12
  Measured by continuous glucose monitoring (CGM) between week 3-4 and week 11-12
Ketones | Week 1-4, week 9-12
  The difference in ketone levels between week 1-4 and week 9-12
Ketoacidosis | Week 1-4, week 9-12
  Occurence of ketoacidosis during the study period and differences between week 1-4 and week 9-12

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, PhD, Principal Investigator — NU Hospital Organization/University of Gothenburg
Locations (1):
- NU Hospital Organization, Uddevalla, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sterner Isaksson S, Olafsdottir AF, Lind M. Design of a randomized cross-over study evaluating effects of carbohydrate intake on glycemic control in persons with type 1 diabetes. Front Nutr. 2023 Mar 13;10:1114317. doi: 10.3389/fnut.2023.1114317. eCollection 2023. PMID 36992911